CLINICAL TRIAL: NCT02357355
Title: Driving Ability in Patients With CMT 1A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jerath U Nivedita (Other)
Responsible Party: Sponsor-Investigator, Jerath U Nivedita, PI, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201307807
Record Dates: First submitted 2015-01-13; First posted 2015-02-06 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: CMT 1A
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMT 1A Group (Active Comparator): Patients with CMT 1A will undergo a driving simulation study. The intervention will be the SIREN driving simulator.
  Interventions: Device: UIHC Driving Simulator
- Control Group (Active Comparator): Patients without CMT 1A who are our normal controls will undergo a driving simulation study. The intervention will be the SIREN driving simulator.
  Interventions: Device: UIHC Driving Simulator

INTERVENTIONS:
Device: UIHC Driving Simulator — This is a driving simulator located in the basement of the hospital. A car will be facing a large video screen of a driving simulation.
  Other Names: SIREN Driving Simulator

SUMMARY:
Charcot Marie Tooth 1A (CMT 1A) is a common inherited disorder of the nerves in the body. The disease can result in difficulties with strength and balance as well as in foot deformities such as high arches, hammer toes, and tight ankles. Because of these difficulties, the disease may affect driving, especially because driving requires quick responses at times such as slamming on the brakes or turning the steering wheel quickly. The following study determines driving performance in individuals who have CMT 1A.

DETAILED DESCRIPTION:
Individuals with CMT 1A will drive in a driving simulator, which involves a car located in a room in the University of Iowa Hospitals and Clinics (UIHC). Individuals will drive in the car as if they are driving in real life and the whole experience is like playing a car video game with a big animated screen. The driving results will be compared to similar aged patients who don't have CMT 1A and have also taken the driving test. If patients with CMT 1A do have driving difficulties compared to those who do not have CMT 1A, the results of the study will try to help patients with CMT1A drive better by ultimately creating devices that might help them use the steering wheel or brake pedal in a safer way.

ELIGIBILITY:
Inclusion Criteria:

* Have CMT 1A
* Have a valid driver's license

Exclusion criteria:

* History of other types of neuropathy (other than CMT 1A)
* History of blindness, seizures, or stroke, dementia/cognitive dysfunction

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Driving Error Rate | 1 year

SECONDARY OUTCOMES:
Deceleration speed | 1 year
Time to braking | 1 year
Time to apply steering maneuvers | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nivedita U. Jerath, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States